CLINICAL TRIAL: NCT05076162
Title: Evaluation of the Relationship Between Vitamin D Level and Emergence Delirium in Children Undergoing Tonsillectomy and/or Adenoidectomy
Brief Title: Vitamin D Level and Emergence Delirium in Children
Status: Completed | Type: Observational
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, SİNAN YILMAZ, Associate Professor, Aydin Adnan Menderes University
Other Study IDs: PAED
Record Dates: First submitted 2021-09-30; First posted 2021-10-13 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-09

CONDITIONS: Delirium
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Serum 25(OH)D levels <12 ng/ml
  Interventions: Diagnostic Test: PAED
- Group 2: Serum 25(OH)D levels ≥12 ng/ml
  Interventions: Diagnostic Test: PAED

INTERVENTIONS:
Diagnostic Test: PAED — Delirium positive or negative

SUMMARY:
In our study, we aimed to evaluate the relationship between vitamin D levels and postoperative delirium in children who had undergone tonsillectomy and/or adenoidectomy.

DETAILED DESCRIPTION:
Patients are assigned to one of two groups. Serum 25(OH)D level will be determined as <12 ng/ml group 1, group 2 with ≥12 ng/ml. ASA I-II children aged 2-10 years who will undergo adenoidectomy and/or tonsillectomy surgery under general anesthesia will be included in the study. In the operating room, the patient will monitored using electrocardiography, pulse oximetry, noninvasive blood pressure measurements, capnography. Under anesthesia, blood samples were taken for serum 25(OH)D levels. After extubation, patients will be taken to the recovery room. Delirium will be evaluated using the PAED (Pediatric Anesthesia Emergence Delirium) scale at 10-minute intervals in the recovery unit. In our study, 25(OH)D level was measured.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status I and II Tonsillectomy and/or Adenoidectomy Surgery

Exclusion Criteria:

* psychological disorders
* emotional disorders
* abnormal cognitive development
* developmental delay
* allergy to the drugs in our protocol

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This was a prospective, single-center, double-blind, randomized study. The primary outcome was the presence or absence of presenting delirium with or without vitamin d deficiency.
  Secondary outcomes, postoperative additional need analgesia. Children aged 2-10 years, ASA (American Society of Anesthesiologists) physical I or II scheduled for tonsillectomy were eligible, with or without adenoidectomy.
Sampling Method: Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
The scale of emergence delirium | up to 30 minutes after arrival in postanesthetic care unit
  After extubation, when spontaneous eye opening and extremity movement started, the patients were taken to the recovery room.
  The patients were evaluated with PAED (Pediatric Anesthesia Emergence Delirium) in the recovery unit. PAED scores were recorded at the time of admission to the postoperative recovery unit and at 10-minute intervals. Patients with a PAED score of 10 and above in any measurement during this time period were recorded as delirium positive.

CONTACTS AND LOCATIONS:
Overall Officials: Sinan Yılmaz, Principal Investigator — institutional affiliation
Locations (1):
- Aydın Adnan Menderes University Faculty of Medicine, Department of Anesthesiology and Reanimation, Aydin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided